CLINICAL TRIAL: NCT01295346
Title: Biomarkers of Mild and Moderate Traumatic Brain Injury
Status: Completed | Type: Observational
Sponsor: Banyan Biomarkers, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: ATO-04b
Record Dates: First submitted 2011-02-07; First posted 2011-02-14 (Estimated); Last update posted 2017-08-08 (Actual); Status verified 2017-08

CONDITIONS: Brain Injuries, Traumatic
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood, serum, plasma
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Traumatic Brain Injury: Patients who present to the health care facility with mild or moderate traumatic brain injury (Glasgow Coma Scale 9-15) within 4 hours of injury
  Interventions: Other: Head CT scan and blood draw

INTERVENTIONS:
Other: Head CT scan and blood draw

SUMMARY:
The purpose of this study is to assess if putative brain injury biomarkers have utility as blood-based traumatic brain injury (TBI) diagnostic and monitoring tools. This will be accomplished by examining the relationships between potential serum-based TBI biomarkers and clinical measures of injury severity, occurrence of complications, and outcome, in subjects with mild or moderate TBI. The assay will be evaluated in a sample population of subjects over the age of 18 who have been referred to the health care provider for closed head injury evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and no more than 80 years of age.
2. Closed injury to the head within 4 hours from symptom onset.
3. Glasgow Coma Scale (GCS) Score of 9-15.
4. Head Computerized Tomography (CT) performed as part of routine care.
5. Subject is willing to undergo the Informed Consent process prior to enrollment.
6. Based upon the Principal Investigator's opinion, subject is an appropriate candidate for the study.

Exclusion Criteria:

1. Participating in another clinical study that may affect the results of either study.
2. Time of injury cannot be determined.
3. Head CT not done as part of clinical emergency care.
4. Primary diagnosis of ischemic or hemorrhagic infarct.
5. Not available for 35 day follow-up visit.
6. Venipuncture not feasible.
7. Blood donation within 1 week of screening.
8. The Subject is otherwise determined by the Investigator to be medically unsuitable for participation in this study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who present to the health care facility with Traumatic Brain Injury (GCS 9-15) within 4 hours of injury.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Assessment of putative TBI markers relative to diagnosis | within 24 hours and at Day 35

SECONDARY OUTCOMES:
Assessment of correlation between putative TBI marker levels and severity of TBI and neuropsychological outcome (per RPQ and ImPACT) | within 24 hours and at Day 35

OTHER OUTCOMES:
Assessment of pituitary status and determination of the presence of autoantibodies | Day 35

CONTACTS AND LOCATIONS:
Overall Officials: Jackson Streeter, MD, Study Chair — Banyan Biomarkers
Locations (7):
- United States (5):
  - Shands at University Florida Gainesville, Gainesville, Florida
  - Dekalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Wayne State University, Detroit, Michigan
  - Washington University, St Louis, Missouri
- Hungary (2):
  - University of Pecs, Pécs
  - University of Szeged, Szeged

REFERENCES:
- [Result] Welch RD, Ayaz SI, Lewis LM, Unden J, Chen JY, Mika VH, Saville B, Tyndall JA, Nash M, Buki A, Barzo P, Hack D, Tortella FC, Schmid K, Hayes RL, Vossough A, Sweriduk ST, Bazarian JJ. Ability of Serum Glial Fibrillary Acidic Protein, Ubiquitin C-Terminal Hydrolase-L1, and S100B To Differentiate Normal and Abnormal Head Computed Tomography Findings in Patients with Suspected Mild or Moderate Traumatic Brain Injury. J Neurotrauma. 2016 Jan 15;33(2):203-14. doi: 10.1089/neu.2015.4149. Epub 2015 Dec 18. PMID 26467555